CLINICAL TRIAL: NCT04323085
Title: Speech-in-Noise Treatments to Improve Hypophonia in Everyday Social Contexts for Individuals With Parkinson's Disease
Brief Title: Speech-in-Noise Treatments for Hypophonia in Parkinson's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Scott Adams, Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 115713
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease; Speech Disorders
Keywords: Hypophonia
MeSH Terms: conditions — Parkinson Disease; Speech Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Speech-in-Noise Treatment Program (Active Comparator): A behavioural speech therapy program involving 12, one-hour treatment sessions over a 4-week period
  Interventions: Behavioral: Speech-in-Noise Treatment Program
- Speech-to-Noise Feedback Device Program (Active Comparator): A speech treatment program involving the use of a speech-to-noise feedback device during 12, one-hour treatment sessions over a 4-week period
  Interventions: Behavioral: Speech-to-Noise Feedback Device Program
- Delayed Treatment (No Intervention): Assessments but no intervention for a period of 13 weeks.

INTERVENTIONS:
Behavioral: Speech-in-Noise Treatment Program — Speech therapy program for hypophonia.
  Arms: Speech-in-Noise Treatment Program
Behavioral: Speech-to-Noise Feedback Device Program — Speech Feedback device program for hypophonia.
  Arms: Speech-to-Noise Feedback Device Program

SUMMARY:
Hypophonia, or reduced speech intensity, is the most prevalent speech symptom in Parkinson's disease (PD) and often leads to significant difficulty communicating in most social situations. Behavioural treatments for hypophonia can be temporarily effective but many individuals fail to retain and transfer improvements beyond the context of the speech clinic. The present study will address the transfer of treatment problem using two new treatment programs. Both treatments focus on improving speech intensity during conversations in different social contexts and a wide range of background noise conditions. The Speech-in-Noise (SIN) treatment program involves training higher speech intensity during variable levels of background noise while receiving real-time intensity feedback from a speech therapist. The second treatment, the Speech-to-Noise Feedback (SNF) device treatment program, involves using a wearable SNF device to provide feedback about an ideal target speech-to-noise level in a wide range of background noise conditions. Forty individuals with PD and their communication partners (i.e. spouse) will be randomly assigned to one of the two treatment programs. To evaluate the effectiveness of the treatments, a wearable recording device will measure daily conversational speech intensity and background noise for 7 consecutive days before, 1 week after, and 12 weeks after treatment.

DETAILED DESCRIPTION:
Parkinson's disease is one of the most common neurodegenerative diseases and is associated with several disabling motor and non-motor symptoms. About 70% of individuals with PD will develop speech impairments. Hypophonia, or reduced speech intensity, is the most prevalent speech symptom and often leads to significant difficulty communicating in most social situations. Behavioural treatments for hypophonia can be temporarily effective but many individuals fail to retain and transfer improvements beyond the context of the speech clinic. These transfer difficulties may be related to cognitive and sensorimotor deficits associated with PD that inhibit the incorporation of new speech strategies into habitual speech. This transfer of treatment problem is a longstanding and major concern in the treatment of speech in PD.

The present study will address the transfer of treatment problem using two new treatment programs. Both treatments focus on improving speech intensity during conversations in different social contexts and a wide range of background noise conditions. The Speech-in-Noise (SIN) treatment program involves training higher speech intensity during variable levels of background noise while receiving real-time intensity feedback from a speech therapist in social situations inside and outside of the clinic. The second treatment, the Speech-to-Noise Feedback (SNF) device treatment program, involves using a wearable SNF device to provide feedback about an ideal target speech-to-noise level in a wide range of background noise conditions inside and outside of the speech clinic.

Forty individuals with PD and their communication partners (i.e. spouse) will be randomly assigned to one of the two treatment programs. In addition, half of the participants will be randomly assigned to a 13-week delayed treatment group and serve as both untreated controls and treated participants.

To evaluate the effectiveness of the treatments, measures of improvement in speech intensity and speech-to-noise levels will be obtained during everyday social conversations. A wearable recording device will measure daily conversational speech intensity and background noise for 7 consecutive days at three time points: before, 1 week after, and 12 weeks after treatment. The effectiveness of treatment will be also measured using two questionnaires and standard, lab-based speech assessments.

It is anticipated that the evaluation and comparison of these two novel treatment paradigms will advance our understanding of procedures that are most effective for enhancing the transfer of treatment for hypophonia into everyday social conversations in individuals with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic PD and hypophonia by a neurologist at least 6 months prior to participation.
* Stabilized on antiparkinsonian medication.
* Good general health.
* 45-85 years old.
* Pass a 50 dB hearing screening and cognitive screening (>20/30 on MOCA).
* Proficient enough in English to participate in speech testing.

Exclusion Criteria:

* History of stroke or an additional neurological or motor control disorder.
* History of speech impairment that is unrelated to PD.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
speech-to-noise ratio | 7 days
  Average speech-to-noise ratio obtained from long-term conversation samples

SECONDARY OUTCOMES:
communication effectiveness ratings | 7 days
  Self-ratings of communication effectiveness using an 8-item questionnaire.
communication participation ratings | 7 days
  Self-ratings of communication participation using a 28 item questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Adams, Principal Investigator — Western University
Locations (1):
- LawsonHRI, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No